CLINICAL TRIAL: NCT01923415
Title: Cross-Sectional Study in Subjects With Active Cutaneous Lupus Erythematosus
Brief Title: A Non-drug Study Profiling Cutaneous Lupus
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR101971; 2013-001531-46 (EudraCT Number); NOCOMPOUNDLUN0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-08-12; First posted 2013-08-15 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic; Lupus Erythematosus, Discoid
Keywords: Lupus Erythematosus, Subacute, Cutaneous; Lupus Erythematosus, Systemic; Lupus Erythematosus, Discoid; Active Cutaneous Lupus Erythematosus; Systemic Cutaneous Lupus Erythematosus; Skin Biopsy; Lesions
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic; Lupus Erythematosus, Discoid | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood from participants with discoid lupus erythematosus (DLE), subacute cutaneous lupus erythematosus (SCLE), and active systemic lupus erythematosus (SLE) with cutaneous involvement.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: SLE: >=10 participants with systemic lupus erythematosus (SLE)
  Interventions: Procedure: No intervention, skin biopsy; Procedure: No intervention, blood collection; Procedure: No intervention, urine collection
- Group 2: DLE: >=10 participants with discoid lupus erythematosus (DLE)
  Interventions: Procedure: No intervention, skin biopsy; Procedure: No intervention, blood collection; Procedure: No intervention, urine collection
- Group 3: SCLE: >=10 participants with subacute cutaneous lupus erythematosus (SCLE)
  Interventions: Procedure: No intervention, skin biopsy; Procedure: No intervention, blood collection; Procedure: No intervention, urine collection

INTERVENTIONS:
Procedure: No intervention, skin biopsy — All participants will have 2 adjacent 4 mm punch biopsies collected from uninvolved and involved skin (a total of 4 biopsies).
Procedure: No intervention, blood collection — Blood for serum analyses will be taken from all participants, blood for DNA analysis only from subjects who consent to this separately.
Procedure: No intervention, urine collection — Urine will be collected from all participants.

SUMMARY:
The purpose of this study is to characterize the clinical and molecular profiles of patients with cutaneous lupus.

DETAILED DESCRIPTION:
This is a Phase 0, multiple-center observational study of biomarkers and clinical parameters in patients with lupus, including discoid lupus erythematosus (DLE), subacute cutaneous LE (SCLE) and active systemic lupus erythematosus (SLE). There is no study-related therapeutic intervention and this protocol will not restrict or introduce any medical interventions including medications. Study participants will undergo procedures that include collection of urine, blood samples, and skin biopsy. At least 30 participants (≥10 DLE, ≥10 SCLE, and ≥10 SLE) will be enrolled in this study. All participants will continue to be managed by their personal physicians per their standard of care. The data obtained in this study will help in the evaluation of new therapeutics for lupus and may facilitate lupus drug discovery. A blood sample for genomic analysis will be collected for research purposes from patients who provide consent and where local regulations permit. There will be a single sample collection time point for each patient. The safety assessments will include laboratory measurements (serum chemistry and hematology), monitoring of adverse events (AEs) related to study procedures, and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* have active DLE or active SCLE confirmed by histological analysis
* have a confirmed diagnosis of SLE with SLE Disease Activity Index (SLEDAI) of >6 and current or historical positive ANA or anti-dsDNA
* have an active skin lesion that can be biopsied
* if using hydroxychloroquine or chloroquine, must be on stable doses for at least 2 months prior to screening.

Exclusion Criteria:

* have an active skin disease other than CLE

  * have any known malignancy within the previous 5 years (with the exception of a non-melanoma skin cancer that has been treated with no evidence of recurrence)
  * have used a topical corticosteroid on active lesion
  * have donated blood (volume >=500 mL) within 56 days prior to screening
  * has been treated with drugs that are associated with CLE induction within 2 months prior to the screening
  * have been treated with >10 mg/day prednisone therapy or equivalent in the last 4 weeks prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants have CLE (either DLE or SCLE) or SLE with cutaneous manifestations
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Assessment of biomarkers in skin biopsies | Day 1
  Investigation of pathways which may be dysregulated in cutaneous lupus lesions.

SECONDARY OUTCOMES:
Urine Biomarkers analysis | Day 1
  The presence of potential biomarkers of disease activity will be explored in urine.
Blood Biomarkers analysis | Day 1
  The presence of potential biomarkers of disease activity will be explored in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Study, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (2):
  - Indianapolis, Indiana
  - Dallas, Texas
- Lodz, Poland